CLINICAL TRIAL: NCT03479632
Title: Aerobic Walking Exercise for Non-Ambulatory Stroke Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00140799
Record Dates: First submitted 2018-03-19; First posted 2018-03-27 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will undergo an aerobic walking program using a treadmill, a body-weight support system, and an assistive device.
  Interventions: Behavioral: Aerobic walking program
- Control Group (Active Comparator): The control group will receive standard physical therapy (PT).
  Interventions: Behavioral: Standard physical therapy

INTERVENTIONS:
Behavioral: Aerobic walking program — Participants will make 24 visits over an 8 week period, having 3 sessions per week. Each session will last about one hour.
  Arms: Intervention Group
Behavioral: Standard physical therapy — Participants will receive standard care they normally would after a stroke.
  Arms: Control Group

SUMMARY:
By doing this study, researchers hope to learn the effects of aerobic exercise on heart, lung, and bone health in people who cannot walk after a stroke.

ELIGIBILITY:
Inclusion Criteria:

* Independent ambulation before stroke
* Be able to understand and follow verbal commands in English
* Have physicians' approval for exercise, and be in stable medical condition
* Participant's first stroke
* Unable to walk independently according to Functional Ambulation Category (FAC) (<2) after in-patient rehabilitation treatment
* Between 6 weeks to 5 years after stroke onset

Exclusion Criteria:

* Current cardiovascular abnormalities other than stroke such as ischemic cardiovascular event or coronary artery bypass surgery less than 3 months ago
* Musculoskeletal disorder which prevents subjects from participating in the exercise
* Resting blood pressure more than 200/110 mm Hg
* Current or previous pulmonary diseases in the past two years
* Osteoporosis and restricted passive movement in the major joints of the lower limbs
* Subjects will be excluded if they are unable to speak or understand English and/or unable to travel to the University of Kansas Medical Center (KUMC) Neuromuscular Research Laboratory

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-03-05 (Actual); Primary Completion 2019-12-05 (Estimated); Study Completion 2020-03-05 (Estimated)

PRIMARY OUTCOMES:
Resting Heart Rate | Change from Baseline to Week 8

SECONDARY OUTCOMES:
Resting blood pressure | Change from Baseline to Week 8
Change in vital capacity (VC) | Change from Baseline to Week 8
Change in forced vital capacity (FVC) | Change from Baseline to Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Wen Liu, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States